CLINICAL TRIAL: NCT06443268
Title: Cerebrovascular Disease: Quality of Life (CODE: QoL)
Acronym: CODE:QoL
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Susanne Wegener, Prof. Dr. med., University of Zurich
Other Study IDs: 2023-00224
Record Dates: First submitted 2024-05-04; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life; Stroke, Acute; Sexual Behavior; Stress; Cortisol Excess; Incontinence, Urinary; Caregiver Burden; Transient Ischemic Attack; Intracerebral Hemorrhage; Cerebrovascular Disorders
Keywords: Stroke, QoL, HRQoL, Patient-Caregiver dyads, Stress, Burden
MeSH Terms: conditions — Stroke; Sexual Behavior; ACTH Syndrome, Ectopic; Urinary Incontinence; Caregiver Burden; Ischemic Attack, Transient; Cerebral Hemorrhage; Cerebrovascular Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hair samples, routine blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with ischemic / hemorrhagic stroke, transient ischemic attack, intracerebral hemorrhage: Patients with ischemic / hemorrhagic stroke, transient ischemic attack, intracerebral hemorrhage
  Interventions: Diagnostic Test: questionnaire, hair samples, blood samples, clinical exam
- Caregivers of patients described above: Caregivers of patients with ischemic / hemorrhagic stroke, transient ischemic attack, intracerebral hemorrhage
  Interventions: Diagnostic Test: questionnaire, hair samples, blood samples, clinical exam
- Patients WITHOUT ischemic / hemorrhagic stroke, transient ischemic attack, intracerebral hemorrhage: Patients WITHOUT ischemic / hemorrhagic stroke, transient ischemic attack, intracerebral hemorrhage or with an event > 3 years ago AND no disability
  Interventions: Diagnostic Test: questionnaire, hair samples, blood samples, clinical exam
- Caregivers of patients above: may include close relatives
  Interventions: Diagnostic Test: questionnaire, hair samples, blood samples, clinical exam

INTERVENTIONS:
Diagnostic Test: questionnaire, hair samples, blood samples, clinical exam — The following parameters will be sequentially assessed in caregivers and patients (baseline, at 3 months and at 12 months): 1) quality of life / functioning will be determined through questionnaires (SF-36, EQ-5DL, ECOG (Eastern Cooperative Oncology Group) / Karnofsky, Barthel Index, ICIQ) 2) stress levels & anxiety levels, caregiver burden will be assessed by the following questionnaires: Distress Thermometer, SBQ-G, GAD-7, PHQ-9, PSS-10, ZBI, PAC. Cortisol will be measured in hair to indicate stress within the past 3 months [18]. Fasting glucose, lipid profiles and HbA1c along with blood count, sodium, potassium, creatinine, TSH (thyroid-stimulating hormone) will be measured in routine blood samples from patients at the time of clinical checkups. Blood pressure, pulse and BMI will be determined during clinical visit in patients and additionally in caregivers.

SUMMARY:
The goal of this observational study is to learn about quality of life, stress and caregiver burden in patients with stroke and their caregivers.

The main question is:

• to discover the factors associated with quality of life and stress in patient-caregiver dyads.

Participants will be asked to fill out questionnaires and agree to provide a hair sample (in order to measure stress hormones in hair) and consent to use of their routine clinical and laboratory data.

Researchers will compare a group of participants without stroke to establish a comparable baseline.

DETAILED DESCRIPTION:
Introduction/Background

In Switzerland, approximately 21,000 people suffer a stroke each year. Stroke causes neurological impairments for those affected and brings about a sudden change in their life situation. The relatives of stroke patients receive new social roles and are challenged in a new way by the morbidity of the affected person, leading to a change in their quality of life and aggravation of stress. Unlike chronic diseases, a stroke occurs suddenly, so relatives have no opportunity to gradually adapt to the new living circumstances or to deal with the new psychosocial roles and demands beforehand. To what extent the daily life of patients and their relatives changes and what impact this has on their quality of life and stress has not been systematically investigated in Switzerland thus far.

Aims and significance of the project

The aim of the project is to systematically assess the quality of life and stress, as well as to capture stress biomarkers in stroke patients and their relatives. The investigators plan to conduct sequential measurements of quality of life and stress hormones at multiple time points over 12 months. The goal is in particular to uncover the relationships between the extent of patients' impairments, their quality of life, and stress in affected individuals and their relatives. This is a first-time project with the goal of learning more about stressors and biological relationships. This will create the basis for a multimodal intervention to improve the quality of life of those affected and their relatives, which will be investigated in a follow-up project.

Methods

The Investigators plan a prospective study with a survey of stroke patients and their relatives regarding their quality of life in everyday life. It will also be examined, how multiple stress biomarkers (which will be determined in blood and hair) are related to quality of life and stress and which clinical factors have a positive and negative influence on the well-being of patients and their relatives.

ELIGIBILITY:
Control group:

Inclusion criteria:

* over 18 years old
* No previous stroke OR previous stroke >3 years ago
* No significant disability (maximum mRS 1)
* ambulatory patients at the University Hospital of Zurich (USZ), Dept. of Neurology
* Patients' AND caregiver's ability to give informed consent
* Patients' AND close relative's / caregiver's willingness to participate

Exclusion criteria:

• Medication with steroid hormones (prednisone, prednisolone, dexamethasone, methylprednisolone, hydrocortisone etc.) within last 3 months

Main Group:

Inclusion criteria:

* over 18 years old
* Patients diagnosed with either transient ischemic attack, ischemic stroke or intracerebral hemorrhage and their caregivers
* Caregiver of a patient as described above, age over 18 years
* Hospitalized or ambulatory patients at the University Hospital of Zurich (USZ) included within 28 days from event.
* Patients' AND caregiver's ability to give informed consent
* Patients' AND caregiver's willingness to participate

Exclusion criteria:

• Medication with steroid hormones (prednisone, prednisolone, dexamethasone, methylprednisolone, hydrocortisone etc.) within last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control group:
  We will include 40 patients without previous stroke OR patients with a minor stroke > 3 years ago and no sustained significant disability (mRS 0 or 1) along with their close relative (to simulate informal caregivers) (total 80 participants).
  Main group:
  We will include 300 patients and informal caregivers with a first cerebrovascular event treated at our clinic > 18 years. The caregivers will be defined as the closest person to the patient with the most contact. (total 600 participants)
Sampling Method: Probability Sample
Enrollment: 680 (Estimated)
Dates: Start 2023-05-27 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life as assessed via Short Form - 36 (SF-36) | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using Short Form - 36 (SF-36)
  Multi-item scale with 8 domains assessing health related quality of life:
  * limitations in physical activities
  * limitations in social activities
  * limitations in usual role activities because
  * pain
  * limitations in social role activities
  * vitality
  * overall mental health
  * overall health
  Domains are scored seperately; Values span from 0 to 100, higher values indicate fewer limitations

SECONDARY OUTCOMES:
Stress | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  as assessed using Perceived Stress Scale - 10 (PSS-10)
  Scoring is based on 2 subscales:
  Subscale 1: Perceived self-efficacy (PSE), range: (4-20)
  Subscale 2: Perceived helplessness (PH), range: (6-30)
  Total score PSS-10 is evaluated by adding both sub scale scores.
  Values span from 10 to 50, higher values indicate higher levels of stress
Positive Aspects of Caregiving: | caregivers at 0, 3 and 12 months after cerebrovascular event.
  Measure of caregiver burden
  Questionnaire: 11 items / Likert scales (1-5)
  Values span from 11 to 55, higher values indicate positive aspects of caregiving
Zarit Burden Interview: | caregivers at 0, 3 and 12 months after cerebrovascular event.
  Measure of caregiver burden
  22 items / Likert scales (0-4) Values span from 0 to 88, higher values indicate higher caregiver burden
Stroke Related Quality of Life | patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using Stroke Impact Scale 3.0 (SIS-3.0)
  SIS-3.0 includes 60 items and assesses 9 domains using Likert scales:
  * Strength - 4 items
  * Hand function - 5 items
  * Activities of daily living - 10 items
  * Mobility - 9 items
  * Communication - 7 items
  * Emotion - 9 items
  * Memory and thinking - 7 items
  * Participation/Role function - 8 items
  * Perceived recovery since stroke onset - single-item VAS (visual analog scale)
  Domains are scored seperately; Values span from 0 to 100, higher values indicate fewer limitations
Anxiety | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using General Anxiety Disorder- (GAD-7)
  7 items / Likert scales (0-3) Values span from 0 to 21, higher values indicate higher level of anxiety and functional impairment
Depression | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using Patient Health Questionnaire - 9 (PHQ-9)
  9 items, evaluated by likert scale (0-3) Values span from 0 to 27, higher values indicate higher probability of depression and decreased functional status
Sexual Quality of Life | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using Sexual Behavior Questionnaire German (SBQ-G)
  Equal base questions (1-6) and gender specific questions m(7-11), f(7-10)
  Single item evaluation with two answer categories
  (0-1) dysfunctional (2-3) functional
  Evaluation of MGISD (Mean Global Index of sexual Dysfunction): Arithmetic mean of 1,4,5,6,8f/11m
Incontinence | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using International Consultation on Incontinence Questionnaire (ICIQ)
  3 Questions regarding urinary incontinence
  * Frequency?
  * Severity?
  * Impact on quality of life?
  Score is sum of answer values (1 + 2 + 3); Range: 0-21
  Scoring Categories
  * slight (1-5)
  * moderate (6-12)
  * severe (13-18)
  * very severe (19-21)
neurological functioning of the patients (NIHSS) | patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using National Institutes of Health Stroke Scale (NIHSS)
  NIHSS
  * 13 assessed functional domains
  * Range 0-42, higher score indicates severe impairment
neurological functioning of the patients (mRS) | patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using modified Rankin Scale (mRS)
  mRS
  • Range: (0-6) 0 = no symptoms, 6 = death, higher score indicates severe impairment
neurological functioning of the patients (Barthel Index) | patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using Barthel Index
  Barthel Index
  * Physical impairment in daily life / self-care
  * score ranges from 0-100
  * higher score indicates fewer limitations
Distress | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using Distress Thermometer
  Assessment with Visual Analog Scale (0-10), higher scale indicates more distress.
  Selection of aspects in life causing distress
Quality of Life (short) | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using EuroQol-5 (EQ5-DL)
  Evaluation of 5 different aspects of health with likert scale (1-5)
  * MOBILITY
  * SELF-CARE
  * USUAL ACTIVITIES
  * PAIN / DISCOMFORT
  * ANXIETY / DEPRESSION
  Each domain is scored individually, higher values indicate higher impairment of quality of life
Quality of Life (short) | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  will be assessed using EuroQol-5 (EQ5-DL)
  Visual analog scale:
  EQ VAS 0-100, higher score indicates better perceived current health
cortisol / cortisone in hair (pg/mg) | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  Stress biomarkers
fasting glucose (mmol/l) | patients at 0, 3 and 12 months after cerebrovascular event.
  Stress biomarkers
HbA1c (in %) | patients at 0, 3 and 12 months after cerebrovascular event.
  Stress biomarkers
Lipid profiles (LDL, HDL, triglycerides in mmol/l) | patients at 0, 3 and 12 months after cerebrovascular event.
  Stress biomarkers
TSH (mU/l) | patients at 0, 3 and 12 months after cerebrovascular event.
  Stress biomarkers
Blood pressure (systolic & diastolic in mmHg) | caregivers and patients at 0, 3 and 12 months after cerebrovascular event.
  Stress biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Wegener, MD, Principal Investigator — University of Zurich
Locations (1):
- Department of Neurology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
not planned at the time of register entry

REFERENCES:
- [Background] Bundesamt für Statistik. Herz und Kreislauf Erkrankungen [online; visited: 21.11.2022] https://www.bfs.admin.ch/bfs/de/home/statistiken/gesundheit/gesundheitszustand/krankheiten/herz-kreislauf-erkrankungen.html
- [Background] Costa TF, Gomes TM, Viana LR, Martins KP, Costa KN. Stroke: patient characteristics and quality of life of caregivers. Rev Bras Enferm. 2016 Sep-Oct;69(5):933-939. doi: 10.1590/0034-7167-2015-0064. English, Portuguese. PMID 27783737
- [Background] Zhang J, Lee DT. Meaning in stroke family caregiving: A literature review. Geriatr Nurs. 2017 Jan-Feb;38(1):48-56. doi: 10.1016/j.gerinurse.2016.07.005. Epub 2016 Sep 23. PMID 27671537
- [Background] Jeong YG, Myong JP, Koo JW. The modifying role of caregiver burden on predictors of quality of life of caregivers of hospitalized chronic stroke patients. Disabil Health J. 2015 Oct;8(4):619-25. doi: 10.1016/j.dhjo.2015.05.005. Epub 2015 May 29. PMID 26123859
- [Background] Haley WE, Roth DL, Hovater M, Clay OJ. Long-term impact of stroke on family caregiver well-being: a population-based case-control study. Neurology. 2015 Mar 31;84(13):1323-9. doi: 10.1212/WNL.0000000000001418. Epub 2015 Mar 4. PMID 25740862
- [Background] Hansel M, Steigmiller K, Luft AR, Gebhard C, Held U, Wegener S. Neurovascular disease in Switzerland: 10-year trends show non-traditional risk factors on the rise and higher exposure in women. Eur J Neurol. 2022 Sep;29(9):2851-2860. doi: 10.1111/ene.15434. Epub 2022 Jun 22. PMID 35661347
- [Background] Schmick A, Juergensen M, Rohde V, Katalinic A, Waldmann A. Assessing health-related quality of life in urology - a survey of 4500 German urologists. BMC Urol. 2017 Jun 19;17(1):46. doi: 10.1186/s12894-017-0235-1. PMID 28629351
- [Background] Hamann J, Herzog L, Wehrli C, Dobrocky T, Bink A, Piccirelli M, Panos L, Kaesmacher J, Fischer U, Stippich C, Luft AR, Gralla J, Arnold M, Wiest R, Sick B, Wegener S. Machine-learning-based outcome prediction in stroke patients with middle cerebral artery-M1 occlusions and early thrombectomy. Eur J Neurol. 2021 Apr;28(4):1234-1243. doi: 10.1111/ene.14651. Epub 2020 Dec 21. PMID 33220140
- [Background] Brott T, Adams HP Jr, Olinger CP, Marler JR, Barsan WG, Biller J, Spilker J, Holleran R, Eberle R, Hertzberg V, et al. Measurements of acute cerebral infarction: a clinical examination scale. Stroke. 1989 Jul;20(7):864-70. doi: 10.1161/01.str.20.7.864. PMID 2749846
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Muller MJ. Development and retest reliability of a German version of the Sexual Behaviour Questionnaire (SBQ-G). Arch Androl. 2007 Mar-Apr;53(2):67-9. doi: 10.1080/01485010600915186. PMID 17453683
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Reis D, Lehr D, Heber E, Ebert DD. The German Version of the Perceived Stress Scale (PSS-10): Evaluation of Dimensionality, Validity, and Measurement Invariance With Exploratory and Confirmatory Bifactor Modeling. Assessment. 2019 Oct;26(7):1246-1259. doi: 10.1177/1073191117715731. Epub 2017 Jun 18. PMID 28627220
- [Background] Ma X, Zhang J, Zhong W, Shu C, Wang F, Wen J, Zhou M, Sang Y, Jiang Y, Liu L. The diagnostic role of a short screening tool--the distress thermometer: a meta-analysis. Support Care Cancer. 2014 Jul;22(7):1741-55. doi: 10.1007/s00520-014-2143-1. Epub 2014 Feb 8. PMID 24510195
- [Background] Bullinger M. German translation and psychometric testing of the SF-36 Health Survey: preliminary results from the IQOLA Project. International Quality of Life Assessment. Soc Sci Med. 1995 Nov;41(10):1359-66. doi: 10.1016/0277-9536(95)00115-n. PMID 8560303
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Sharpley CF, McFarlane JR, Slominski A. Stress-linked cortisol concentrations in hair: what we know and what we need to know. Rev Neurosci. 2011 Dec 8;23(1):111-21. doi: 10.1515/RNS.2011.058. PMID 22150070
- [Background] Kim JH, Kim O. Influence of mastery and sexual frequency on depression in Korean men after a stroke. J Psychosom Res. 2008 Dec;65(6):565-9. doi: 10.1016/j.jpsychores.2008.06.005. Epub 2008 Oct 28. PMID 19027446
- [Background] Oyewole OO, Ogunlana MO, Gbiri CAO, Oritogun KS. Prevalence and impact of disability and sexual dysfunction on Health-Related Quality of Life of Nigerian stroke survivors. Disabil Rehabil. 2017 Oct;39(20):2081-2086. doi: 10.1080/09638288.2016.1219395. Epub 2016 Aug 22. PMID 27548503
- [Background] Forsberg-Warleby G, Moller A, Blomstrand C. Life satisfaction in spouses of patients with stroke during the first year after stroke. J Rehabil Med. 2004 Jan;36(1):4-11. doi: 10.1080/16501970310015191. PMID 15074432
- [Background] Kjork E, Blomstrand C, Carlsson G, Lundgren-Nilsson A, Gustafsson C. Daily life consequences, cognitive impairment, and fatigue after transient ischemic attack. Acta Neurol Scand. 2016 Feb;133(2):103-110. doi: 10.1111/ane.12435. Epub 2015 May 8. PMID 25955112
- [Background] Hinz A, Klein AM, Brahler E, Glaesmer H, Luck T, Riedel-Heller SG, Wirkner K, Hilbert A. Psychometric evaluation of the Generalized Anxiety Disorder Screener GAD-7, based on a large German general population sample. J Affect Disord. 2017 Mar 1;210:338-344. doi: 10.1016/j.jad.2016.12.012. Epub 2016 Dec 18. PMID 28088111
- [Background] Tarlow, B. J., Wisniewski, S. R., Belle, S. H., Rubert, M., Ory, M. G., & Gallagher-Thompson, D. (2004). Positive Aspects of Caregiving: Contributions of the REACH Project to the Development of New Measures for Alzheimer's Caregiving. Research on Aging, 26(4), 429-453. https://doi.org/10.1177/0164027504264493